CLINICAL TRIAL: NCT02869737
Title: Utility of Point-of-care Device for Rapid Determination of Cogulopathy in Trauma Patients
Acronym: Coaguchek
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: CECIC 2015-03
Record Dates: First submitted 2016-08-09; First posted 2016-08-17 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Severe Trauma
Keywords: Point of Care Device; post traumatic coagulopathy
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Coagucheck, Roche, France — Capillary puncture for POC INR measurement

SUMMARY:
Traumatic coagulopathy is frequent and is an independent risk factor of mortality. Its detection mainly relies upon classic biological test like the prothrombin time and the international normaliezd ratio (INR). These tests are not available at the bedside. Point of care (POC) device for INR measurement are now available like the Coaguchek, Roche, France. The aim of the present study is to test the correlation between the POC INR and the laboratory INR.

ELIGIBILITY:
Inclusion Criteria:

* Age > 15 y-o
* Admission for severe trauma

Exclusion Criteria:

* Patients under oral anticoagulant

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admited for a suspicion of severe trauma wirth active bleeding in a level I trauma center
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Concordance between POC INR and laboratory INR using 3 classes: normal < 1.1, moderate : 1.1-1.5, severe: >1.5 | Admission

SECONDARY OUTCOMES:
Prediction of RBC transfusion | 24 hours post admission
Prediction of FFP transfusion | 24 hours post admission
In-hospital mortality assessed using patients' files | up to Day 28
Injury severity (ISS) | Day 1
Organ failure measured with the SOFA score at Day 1 | Day 1

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mistral T, Boue Y, Bosson JL, Manhes P, Greze J, Brun J, Albaladejo P, Payen JF, Bouzat P. Performance of point-of-care international normalized ratio measurement to diagnose trauma-induced coagulopathy. Scand J Trauma Resusc Emerg Med. 2017 Jun 21;25(1):59. doi: 10.1186/s13049-017-0404-y. PMID 28637514